CLINICAL TRIAL: NCT05877521
Title: Adapting Mindfulness-oriented Recovery Enhancement (MORE) for Cancer Pain Relief: The MORE Relief Trial
Brief Title: Mindfulness-oriented Recovery Enhancement (MORE) for Cancer Pain Relief
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-082
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain; Cancer Pain
Keywords: chronic pain; cancer pain; Mindfulness-oriented Recovery Enhancement; MORE; mindfulness-based interventions; MBIs; Memorial Sloan Kettering Cancer Center; 23-082
MeSH Terms: conditions — Chronic Pain; Cancer Pain | interventions — Standard of Care; Pain Management

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wait List Control (WLC) Usual Care Procedure (Placebo Comparator): Participants in the WLC group continue to receive their standard medical care and pain management as prescribed by their physicians or other health care providers.
  Interventions: Other: Standard of Care for Pain Management
- 16-hour MORE treatments (Experimental): Patients in the 16-hour MORE format will receive one 2hrs treatment a week for 8 consecutive weeks (as per study schema: from week 1 to week 8).
  Interventions: Behavioral: MORE treatments
- 8-hour MORE treatments (Experimental): Patients in the 8-hour MORE format will receive one 2hrs treatment a week for 4 consecutive weeks (as per study schema: from week 1 to week 4).
  Interventions: Behavioral: MORE treatments
- 2-hour MORE treatments (Experimental): Patients in the 2-hour MORE format will receive one 2hrs treatment (as per study schema: in week 1).
  Interventions: Behavioral: MORE treatments

INTERVENTIONS:
Behavioral: MORE treatments — MORE participants will also be asked to engage in 15 minutes/day of skill practice at home, and complete daily diaries of mindfulness practice time
  Arms: 16-hour MORE treatments; 2-hour MORE treatments; 8-hour MORE treatments
Other: Standard of Care for Pain Management — Participants in the WLC group continue to receive their standard medical care and pain management as prescribed by their physicians or other health care providers.
  Arms: Wait List Control (WLC) Usual Care Procedure

SUMMARY:
The purpose of this study is to evaluate whether or not mindfulness-based interventions/MBIs may help reduce chronic pain in participants who have cancer-related chronic pain. MBIs are therapeutic programs that use mindfulness meditation practices to help people focus on the present moment, as well as encourage acceptance of thoughts, emotions, and body sensations. The researchers think that an MBI treatment called Mindfulness-oriented Recovery Enhancement (MORE) may help people who are experiencing cancer-related chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age ≥ 18 years or older
* A history of cancer with no restrictions placed on type of cancer
* Determined to be either no-evidence of disease or stable oncological disease by referring or study physicians/advanced practice providers
* Having a pain (musculoskeletal, generalized, or neuropathic) rating of 4 or greater in worst pain on a 0-10 numerical rating scale in the preceding week
* Having had pain for at least 3 months and at least 15 days with pain in the preceding 30 days
* Willing to adhere to all study-related procedures, including randomization to one of two treatment arms: MORE or WLC
* Ability to attend video-call session and a quiet/private location

Exclusion Criteria:

* Active suicidality or schizophrenia
* Plan to initiate palliative radiation or interventional pain procedure within the next 12 weeks
* Cognitive impairment preventing completing PRO independently or participate in virtual MORE as evaluated by study clinicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2027-05-16 (Estimated); Study Completion 2027-05-16 (Estimated)

PRIMARY OUTCOMES:
Rate of participant enrollment to the study | 12 months
  Feasibility of the intervention will be determined by Rate of participant enrollment to the study

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Bryl KL, Hanley AW, Baser RE, Desai K, Dowd M, Li Q, Sandweiss B, Garland EL, Mao JJ. Mindfulness-Oriented Recovery Enhancement for Cancer Pain Relief: Pilot Randomized Controlled Trial. J Pain Symptom Manage. 2026 Jan 3:S0885-3924(25)01035-8. doi: 10.1016/j.jpainsymman.2025.12.024. Online ahead of print. PMID 41490669
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org